CLINICAL TRIAL: NCT07136337
Title: The Diagnostic Utility of T Immunoglobulin G and T Immunoglobulin M Biomarkers in Patients With Systemic Lupus Erythematosus Disease : Associations With Disease Activity and Damage
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mai Hany Ahmed Ibrahim, Mai Hany Ahmed Ibrahim, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: TigG and TigM in SLE
Record Dates: First submitted 2025-08-10; First posted 2025-08-22 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Systemic Lupus Erythematosus
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Systemic lupus erythematosus patients (Experimental): 4 ml. of fresh venous blood will be collected from each patient on EDTA tube and will be used for detection of the following : T cell immunoglobulin G ( TIgG) and T cell immunoglobulin M (TIgM) by flow cytometry
  Interventions: Diagnostic Test: 4 ml. of fresh venous blood will be collected from each patient on EDTA tube and will be used for detection of the following : T cell immunoglobulin G ( TIgG) and T cell immunoglobulin M (TIgM) by
- Helthy control (Other): 4 ml. of fresh venous blood will be collected from each patient on EDTA tube and will be used for detection of the following : T cell immunoglobulin G ( TIgG) and T cell immunoglobulin M (TIgM) by flow cytometry
  Interventions: Diagnostic Test: 4 ml. of fresh venous blood will be collected from each patient on EDTA tube and will be used for detection of the following : T cell immunoglobulin G ( TIgG) and T cell immunoglobulin M (TIgM) by

INTERVENTIONS:
Diagnostic Test: 4 ml. of fresh venous blood will be collected from each patient on EDTA tube and will be used for detection of the following : T cell immunoglobulin G ( TIgG) and T cell immunoglobulin M (TIgM) by — 4 ml. of fresh venous blood will be collected from each patient on EDTA tube and will be used for detection of the following : T cell immunoglobulin G ( TIgG) and T cell immunoglobulin M (TIgM) by flow cytometry

SUMMARY:
The SLE is heterogeneous multisystem autoimmune disease with complex pathogenesis involves multiple cellular components of the innate and adaptive immune systems, presence of autoantibodies and immune complexes, engagement of the complement system, dysregulation of several cytokines including type I interferons, and disruption of the clearance of nucleic acids after cell death(1,2,3).

Among the putative mechanisms leading to the pathogenic breakdown of immune tolerance in SLE is the development of auto reactive T Cells, which contribute to pathologic activation of B cells, dysfunction of regulatory T Cells and aberrant production of pro-inflammatory cytokines (4,5) Autoantibodies targeting the T Cell Receptor (TCR)/CD3 have been demonstrated to activate Ca2+/calmodulin-dependent kinase IV (CaMKIV), resulting in diminished IL-2 production and low serum IL-2 levels are commonly observed in SLE (6,7,8,9) T Cell autoantibodies have been shown to influence T Cell signalling, migration, and adhesion, contributing to organ-specific targeting in SLE. These findings suggest that T Cell autoantibodies are active participants in disease pathogenesis and , supporting their potential as biomarkers for diagnosis and disease activity (10) Delays in SLE diagnosis, often due to the limitations of current biomarkers, can lead to worsened outcomes (11). Improved diagnostic markers, such as the T Cell biomarkers described here, could help reduce these delays , improve patient care and improve the ability of clinicians to differentiate between SLE and patients with falsely positive ANA (12) To the best of our knowledge, only a limited number of studies have explored the role of T cell autoantibodies in diagnosing and monitoring disease activity in SLE (12), and none have examined their association with lupus nephritis and disease damage index .

ELIGIBILITY:
Inclusion Criteria:

* : Adult SLE Patients ( >18 years ) who are fulfilling the 2019 ACR\EULAR classification criteria of systemic lupus erythematosus

Exclusion Criteria:

1. SLE patients <18 years old
2. Patients with other autoimmune diseases (systemic sclerosis , sjogren syndrome, rheumatoid arthritis dermatomyositis, mixed connective tissue disease).
3. Pregnant and lactating women .

   -

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
to measure the level of these novel biomarkers and evaluate their role as diagnostic biomarkers in SLE . | 2 years

SECONDARY OUTCOMES:
Study the correlation of TIgG and TIgM with different SLE manifestations and with disease activity and damage index | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut university hospital, Asyut, Asyut Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related Info — https://www.frontiersin.org/journals/immunology/articles/10.3389/fimmu.2025.1518208/full